CLINICAL TRIAL: NCT05200676
Title: Cardiac Arrhythmias in Greenland
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Nadja Albertsen, Principal Investigator, Aalborg University Hospital
Other Study IDs: KVUG 2020-18
Record Dates: First submitted 2021-12-13; First posted 2022-01-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Arrhythmia; Autonomic Neuropathy
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main group: All included in the study will offered to participate in:
  * ePatch-monitoring
  * Blood pressure measurement
  * Cardial vagal tone
  * Questionnaire-assessment
  Interventions: Device: ePatch
- Subgroup: Part of the study-population will be offered to participate in en examination with a SmartPill. The Smartpill measures pressure, pH, temperature and movement in the gut. These measurements gives an indication of the function of the autonomic nervous system (ANS) of the participant. Although measured in the gut, this is relevant as ANS-dysfunction may cause arrhythmias.
  Only a subgroup of the study population will be offered to participate due to the cost of this examination.
  Interventions: Device: ePatch; Device: SmartPill

INTERVENTIONS:
Device: ePatch — ePatch registers the heart rate continuously when attached to the chest of the participant.
Device: SmartPill — SmartPill is swallowed and passes through the digestive system while sending information to a recording device. The pill is passed in the stool and not reused.
  Groups: Subgroup

SUMMARY:
The study is a phd-study comprising several substudies focusing on cardiac arrhythmias, mainly atrial fibrillation, among Greenlanders in Greenland.

Some previous studies have indicated that the prevalence may be lower than among Westerners, however; studies have also indicated that atrial fibrillation is underdiagnosed.

These studies aim to:

* Estimate the prevalence of AF among Greenlanders in Greenland aged 55 years or older.
* Estimate the prevalence of well-known risk factors among those found to have AF
* Explore the symptoms of those affected by AF in Greenland
* Among part of the participants: estimate the prevalence of autonomic neuropathy as this may cause arrhythmias.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia globally and a major risk factor for ischemic strokes, transient ischemic attacks, increased morbidity and mortality.

Risk factors for AF include diabetes, hyperthyroidism, hypertension, obesity, ischemic heart disease (IHD), age and gender with men generally having a higher risk of developing AF.

The current prevalence of cardiac arrhythmias in Greenland is unknown. From 1962 to 1964 12-lead electrocardiograms (ECGs) were performed on 181 adults and only one of these showed AF. A more recent study from 2013 estimating the incidence of ischemic strokes among Greenlanders found that five percent of this study-population had been diagnosed with AF before the incident, while 32.4 % were diagnosed after the incident, suggesting that AF may be underdiagnosed. Comparing the age of the patients to data from Denmark, the authors found that the incidence rate for stroke was higher among almost all younger age groups in Greenland.

Previous studies have shown that ethnicity may influence the risk of developing AF. The genetic profile of the Greenlandic Inuit has already been shown to have a major impact on the risk of developing type 2 diabetes.

Regarding other AF-related risk factors, hypertension is common with a prevalence of app. 40% among men and 32% among women based on self-reported data, and a study comparing data from ECGs performed in 1963 with more current data has shown a rise in the incidence of IHD.

Furthermore, the number of obese people in Greenland is steadily rising and between 1963 and 2008, the proportion of obese people (BMI≥30) increased from 4.0% to 33.2% for men and 8.3% to 24.5% for women between 50 to 69 years.

In conclusion, the risk factors for cardiac arrhythmias are increasing in Greenland and the overall aim of this study is to estimate the prevalence, risk factors, mortality, morbidity and treatment of arrhythmias in Greenland.

Relevance: as mentioned above, this study aims to estimate the prevalence, risk factors, mortality, morbidity and treatment of arrhythmias in Greenland, all of which is currently unknown. By doing this, the study aims to not only improve the treatment rate of arrhythmias, but also lower the prevalence of diseases such as strokes, which are often caused by arrhythmias. By lowering this prevalence, some deaths and cases of disability can be prevented. Furthermore, the investigators hope to assess whether arrhythmias are influenced differently by ethnicity and risk factors such as diabetes in Greenland than in Europe and if patients with certain diseases and/or symptoms have a higher risk of developing arrhythmias and should be monitored more closely.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years old
* Greenlandic ethnicity based on parents' birth place.
* No history of cardiac disease or arrhythmia

Exclusion Criteria:

* Celiac disease (for the SmartPill-study)

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People aged 50 years or older living in Nuuk at the time of recruitment (January 2022) will be invited to participate. Ethnicity and eligibility will be assessed when contacting potential participants after the written invitation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Prevalence od cardiac arrhythmiaa / atrial fibrillation in the population older than 50 years | Completed within 6 months.
  Whether participant has an arrhythmia or not - and if the participant does, what kind of arrhythmia. ePatch recordings will be analysed by the producing company after the completion of the recordings of all participants.
Prevalence of common symptoms of arrhythmias | Completed within 8 months
  Questionnaire-based. Participants will be asked about the most common symptoms of arrhythmias (palpitations, chest pains, feeling a "loss of a beat", dizziness). Depending on the results, the questionnaires may be followed-up by qualitative interviews. The questionnaires are filled out as part of the trial. Results will be entered into a database (RedCap) continuously and analysed after the trial.
Prevalence of risk factors for AF | Completed within 8 months
  Questionnaire-based. Participants will be asked about common risk factors for AF (family history, smoking, hypertension, ischemic heart disease, thyroid disease, age, gender). The questionnaires are filled out as part of the trial. Results will be entered into a database (RedCap) continuously and analysed after the trial.
Number of patients with ANS-neuropathy | Within 10 months
  Based on the recordings of the SmartPill-system. Data will be analysed externally by the MechSense-group at Aalborg University Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Albertsen, MD, PhD, Principal Investigator — Aalborg University / University of Greenland and Aalborg University Hospital
Locations (1):
- Ilisimatusarfik, Nuuk, Greenland

IPD SHARING:
Plan to Share IPD: No